CLINICAL TRIAL: NCT02632578
Title: A Comparison of Immune Responses to the Licensed Trivalent Inactivated Influenza Vaccine in HIV-positive and HIV-negative Subjects
Brief Title: Influenza Vaccine in HIV Study
Status: Completed | Type: Observational
Sponsor: University of Melbourne (Other)
Responsible Party: Principal Investigator, Prof Stephen Kent, Professor, University of Melbourne
Other Study IDs: Kent001; AISRF08020 (Other Grant/Funding Number: The Australia-India Strategic Research Fund); 1041832, 1042634, 1052979 (Other Grant/Funding Number: The Australian National Health and Medical Research Council)
Record Dates: First submitted 2015-12-14; First posted 2015-12-16 (Estimated); Last update posted 2015-12-16 (Estimated); Status verified 2015-12

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV-positive
  Interventions: Biological: 2015 Fluvax® vaccine, BioCSL (a licensed influenza vaccine)
- HIV-negative
  Interventions: Biological: 2015 Fluvax® vaccine, BioCSL (a licensed influenza vaccine)

INTERVENTIONS:
Biological: 2015 Fluvax® vaccine, BioCSL (a licensed influenza vaccine) — Subjects received licensed influenza vaccine (Fluvax®), 1ml intramuscular injection.

SUMMARY:
The aims of this study are:

1. to investigate if HIV infection alters the antibody responses to influenza and
2. to assess the ability of licensed influenza vaccine to induce functional non-neutralising antibodies in HIV-infected and HIV-uninfected subjects.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive by licensed diagnostic test (for HIV-positive group only)
* Planning to receive the seasonal influenza vaccine outside the study
* Provision of written informed consent

Exclusion Criteria:

* Previous allergy to influenza vaccination
* Pregnancy or planning to become pregnant
* Unwilling or unable to provide blood samples

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects are recruited from two sites in Melbourne, Australia:
  * Melbourne Sexual Health Centre (HIV-positive and HIV-negative subjects)
  * The University of Melbourne at the Peter Doherty Institute for Infection and Immunity (HIV-negative subjects only)
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Anti-influenza antibody responses in plasma with Fc-mediated functions | Four weeks after influenza vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kent, Professor, Principal Investigator — University of Melbourne

IPD SHARING:
Plan to Share IPD: No